CLINICAL TRIAL: NCT02278822
Title: Pilot Study of Oral Liposomal Glutathione Supplementation on Levels of Glutathione in Blood and Biomarkers of Oxidative Stress and Immune Function in Healthy Adults
Brief Title: Oral Liposomal Glutathione Supplementation in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Raghu Sinha, Associate Professor of Biochemistry and Molecular Biology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000405
Record Dates: First submitted 2014-10-11; First posted 2014-10-30 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose oral liposomal glutathione (Experimental): Intervention: low dose oral liposomal glutathione supplementation. 500 mg oral liposomal glutathione each day for 4 weeks.
  Interventions: Other: Low dose oral liposomal glutathione supplementation
- High dose oral liposomal glutathione (Experimental): Intervention: high dose oral liposomal glutathione supplementation. 1000 mg oral liposomal glutathione each day for 4 weeks.
  Interventions: Other: High dose oral liposomal glutathione supplementation

INTERVENTIONS:
Other: Low dose oral liposomal glutathione supplementation — Low dose oral liposomal glutathione supplementation
  Arms: Low dose oral liposomal glutathione
Other: High dose oral liposomal glutathione supplementation — High dose oral liposomal glutathione supplementation
  Arms: High dose oral liposomal glutathione

SUMMARY:
This trial is designed to provide evidence of the efficacy of liposomal glutathione supplementation on healthy adults. The investigators anticipate that liposomal glutathione supplementation will enhance the levels of blood glutathione and improve the immune functions.

DETAILED DESCRIPTION:
This is a randomized study on healthy individuals. The study design includes the recruitment of 12 healthy male and female subjects (50-80 yr of age) randomized into 2 groups of 6 each (liposomal glutathione at 500 mg/day or liposomal glutathione at 1000 mg/day). Blood and urine samples will be obtained from all subjects at baseline. Eligible subjects will be required to have not have taken any high dose antioxidant supplements for at least 1 month prior to the study. Subjects will then begin supplementation according to the following schedule: Group A, liposomal glutathione (500 mg daily), Group B, liposomal glutathione (1000 mg daily)

Eligible participants who sign the informed consent will be randomly assigned to either low dose or high dose glutathione groups. Participants will be asked not to consume any other high-dose vitamin, multi-vitamin, or mineral supplements containing glutathione throughout the study in order to prevent variation in dose of supplemental liposomal glutathione between subjects. Participants are to limit their consumption of alcohol in the study to no more than 5 oz. of alcohol per week. Supplementation will continue for 1 month with biological samples collected at 1, 2 and 4 weeks after baseline.

Levels of glutathione will be measured in whole blood, erythrocytes, lymphocytes and plasma. The biomarkers of oxidative stress will include urinary 8-isoprostane and urinary 8-hydroxydeoxyguanosine. Immune function biomarkers will be analyzed including lymphocyte proliferation and natural killer (NK) cell cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy English-speaking male and female volunteers
* Baseline blood glutathione level of ≤ 0.9 mmol/l
* Non-smoking individuals

Exclusion Criteria:

* No history or evidence of disease including cancer, diabetes, heart disease.
* Not taking glutathione as a dietary supplement
* Not taking high-dose antioxidant supplements

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Glutathione levels in blood | Baseline and 4 weeks

SECONDARY OUTCOMES:
Measure immune function biomarkers in blood | Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raghu Sinha, PhD, Principal Investigator — M.S. Hershey Medical Center
Locations (1):
- M.S. Hershey Medical Center, Hershey, Pennsylvania, United States